CLINICAL TRIAL: NCT05469568
Title: Hybrid Rehabilitation Approach Through Group Exercise and Telerehabilitation in Patients With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hybrid rehabilitation approach
Record Dates: First submitted 2022-06-23; First posted 2022-07-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Telerehabilitation; Circuit Training; Movement Skills; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit training and telerehabilitation (Experimental): The experimental group will participate in a 12-week rehabilitation program, including training once a week. After the end of this outpatient program, participants will gain access to a mobile application in which participants will record all their physical activities.The mobile application will also include a library of exercises taught during the outpatient program so patients can practice them at home.
  Interventions: Other: Circuit training followed by telerehabilitation
- Usual Care (Sham Comparator): Patients have usual care and usual information about importance of regular movement activities and recommendation of proper exercises. Patients don't visit ambulatory rehabilitation program and they don't have access to an application
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Circuit training followed by telerehabilitation — Patients participate in an ambulatory rehabilitation program (12 weeks) and then gain access to mobile application to record their movement activities. This application will aslo inlude a library with exercise vidoes from the ambulatory program. These videos should inspire patients to do the exercises at home.
  Arms: Circuit training and telerehabilitation
Other: Usual care — Patients have usual information about importance of regular movement activities and recommendation of proper exercises
  Arms: Usual Care

SUMMARY:
The aim of the study is to determine the benefits of outpatient group rehabilitation with subsequent telerehabilitation. The patient will participate in a 12-week circuit training, including training once a week in a group of six under the guidance of two physiotherapists. After the outpatient rehabilitation, the patient will gain access to a mobile application and will be asked to record all physical activities there.

DETAILED DESCRIPTION:
In the Czech population more than 20,000 people have been diagnosed with multiple sclerosis (MS), an autoimmune disease affecting a patient's central nervous system. This disease has a wide range of symptoms, with the most common ones being various motor disorders that negatively affect the locomotor function and patients' quality of life.

The positive effect of physical activity on human health is well known. This study aims to examine the effect of hybrid exercise program on people with MS. This exercise program includes ambulatory circuit training for twelve weeks followed by telerehabilitation. The aim of the study is to find out whether the exercise program will positively affect the movement skills of probands and improve their quality of life. Testing will done before the start of the exercise program, after twelve weeks and after 6 months. Movement skills will be tested by a set of movement tests called miniBEST test. For measuring quality of life the investigators will the SF-36 questionnaire will be used. Another goal will analyze participants' satisfaction with the intervention and adherence to regular physical activity.

The investigators anticipate that regular physical training combined with telerehabilitation will increase the motivation and effectiveness of independent training in people with MS leading to improvment of physical fitness, physical activity levels and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmed diagnosis of Multiple Sclerosis based on McDonald criteria
* Minimal one month from last relapse
* Possibility to use smartphone or tablet because of using rehabilitation application

Exclusion Criteria:

* Illnesses which can limiting exercises activities (e.g. orthopedic, cardiology or other neurological diseases)
* Cognitive deficit which can limiting cooperation (fill a questionnaire, comply with movement task, using application)
* Relapse of diseases during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Movement skills score at 12 weeks and 6 months | Baseline, 12 weeks, 6 months
  Mini Balance Evaluation Systems Test (Mini BESTest) - 14-item scale for measure postural stability. Maximum value is 28 points, minimum value is 0 point. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Depression score at 12 weeks and 6 months | Baseline, 12 weeks, 6 months
  Beck's Depression Inventory (BDI) - 21-item, self-report rating. Maximum value is 63 points, minimum value is 0 point. Higher scores mean a worse outcome.
Change from Baseline Walking skills score at 12 weeks and 6 months | Baseline, 12 weeks, 6 months
  12-Item Multiple Sclerosis Walking Scale - self-report rating. Maximum value is 60 points, minimum value is 12 point. Higher scores mean a worse outcome.
Exercise adherence | 6 months
  Number of added movement activities in application. Higher scores mean better adherence to exercise.
Change from Baseline Health related quality of life score at 12 weeks and 6 months | Baseline, 12 weeks, 6 months
  Short Form Survey (SF-36) - 36-item. Maximum value is 100 points, minimum value is 36 point. Higher score mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ladislav Batalik, Principal Investigator — Department of Rehabilitation, University Hospital Brno, Czech Republic
Locations (1):
- Michaela Sládečková, Brno, Czech Republic, Czechia